CLINICAL TRIAL: NCT04144855
Title: A Phase I, Open-label, Multicenter, Dose Escalation and Expansion Study to Evaluate the Tolerance and Pharmacokinetics of TQB3474 Injection
Brief Title: A Study to Evaluate the Tolerance and Pharmacokinetics of TQB3474 Injection
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3474-I-01
Record Dates: First submitted 2019-10-24; First posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3474 injection (Experimental): Participants receive TQB3474 injection by intravenous (IV) infusion on Day 1, 8, 15, 22 of each 28 day cycle.
  Interventions: Drug: TQB3474 injection

INTERVENTIONS:
Drug: TQB3474 injection — This is a kind of heat shock protein (HSP90) inhibitor.

SUMMARY:
This is a study to evaluate the tolerance, dose-limiting toxicity (DLT), phase II recommended dose (RP2D), and maximum tolerated dose (MTD) of single and multiple oral doses of TQB3474 in patients with advanced malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

1.18 and 70 years old.

2. Histologically or cytologically confirmed advanced solid tumors.

3. Has the surgery more than 4 weeks before the first dose.

4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1.

5. Life expectancy ≥12 weeks.

6. Adequate organ system function.

7. Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study.

8. Understood and signed an informed consent form.

Exclusion Criteria:

1. Has received chemotherapy or radiotherapy within 4 weeks before the first dose.
2. Hypersensitivity to TQB3474 or its excipient.
3. Has factors that impact on intravenous infusion of drugs and venous blood collection.
4. Has severe gastrointestinal disease within 4 weeks before the first dose.
5. Has severe eye disease.
6. Breastfeeding or pregnant women.
7. Has brain metastases.
8. HCV antibody and HCV-RNA positive; Syphilis positive; HBsAg positive and HBV DNA positive (≥1000 copies /mL).
9. Has infection that need systemic treatment during screening.
10. Has participated in any other clinical trial within 4 weeks before the first dose.
11. According to the judgement of the researchers, there are other factors that subjects are not suitable for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-11-27 (Actual); Primary Completion 2020-11-27 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Baseline up to 28 days
  Subjects appear the following toxic reaction relate to the drug after treatment within 28 days ：III °or above of non-hematological toxicity, IV° hematological toxicity , III ° neutropenia associated with fever, III ° thrombocytopenia with bleeding.

SECONDARY OUTCOMES:
Cmax | 0hour, 0.5hour, end of infusion, 5minutes, 15minutes, 0.5hour, 1hour, 2hour, 4hour, 7hour, 12hour, 24hour, 48hour, 144hour after infusion of day 1 and day 22; Hour 0, end of infusion of day 8 and day 15, hour 0 of day 29.
  Cmax is the maximum plasma concentration of TQB3474 or metabolite(s).
Tmax | 0hour, 0.5hour, end of infusion, 5minutes, 15minutes, 0.5hour, 1hour, 2hour, 4hour, 7hour, 12hour, 24hour, 48hour, 144hour after infusion of day 1 and day 22; Hour 0, end of infusion of day 8 and day 15, hour 0 of day 29.
  To characterize the pharmacokinetics of TQB3474 by assessment of time to reach maximum plasma concentration.
AUC0-t | 0hour, 0.5hour, end of infusion, 5minutes, 15minutes, 0.5hour, 1hour, 2hour, 4hour, 7hour, 12hour, 24hour, 48hour, 144hour after infusion of day 1 and day 22; Hour 0, end of infusion of day 8 and day 15, hour 0 of day 29.
  To characterize the pharmacokinetics of TQB3474 by assessment of area under the plasma concentration time curve from zero to infinity.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Guizhou Cancer Hospital, Guiyang, Guizhou
  - Yongsheng, Chengdu, Sichuan